CLINICAL TRIAL: NCT00526929
Title: A Pilot Study Evaluating Once Every Other Week Administration of Fixed Doses of Novel Erythropoiesis Stimulating Protein (NESP) to Subjects With Chronic Renal Insufficiency (CRI)
Brief Title: Fixed Dose NESP Study in Subjects With CRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 990151
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2009-05-22 (Estimated); Status verified 2009-05

CONDITIONS: Pre-Dialysis
MeSH Terms: interventions — Darbepoetin alfa

ARMS (1):
- darbepoetin alfa (Experimental): darbepoetin alfa (NESP)
  Interventions: Drug: darbepoetin alfa

INTERVENTIONS:
Drug: darbepoetin alfa — 10 mcg NESP administered SC every other week 15 mcg NESP administered SC every other week 20 mcg NESP administered SC every other week 30 mcg NESP administered SC every other week 40 mcg NESP administered SC every other week 50 mcg NESP administered SC every other week 60 mcg NESP administered SC every other week 80 mcg NESP administered SC every other week 100 mcg NESP administered SC every other week

SUMMARY:
Multicenter, open-label, single-arm, fixed dose study of darbepoetin alfa in subjects with Chronic Renal Insufficiency (CRI). Subjects will be screened for 2 weeks during which time blood will be drawn and vital signs will be taken. Upon enrollment, subjects will receive SC darbepoetin alfa administered once every other week for 24 weeks. Darbepoetin alfa will be titrated in fixed-dose steps to maintain a hemoglobin of 11.0 - 13.0. During the study, laboratory assessments will be completed and vital signs will be taken. Subjects will enter a 1-week post-treatment observation and evaluation period after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age
* CRI with a creatinine clearance of less than 40 mL/min
* Hemoglobin less than 11.0 g/dL
* Serum vitamin B12 and folate levels above the lower limit of normal and iron replete

Exclusion Criteria:

* Received rHuEPO therapy in the last 12 weeks
* Expected to initiate renal replacement therapy within 24 weeks or a recipient of a renal transplant
* Uncontrolled hypertension
* Seizure activity, CHF, hyperparathyroidism, major surgery, HIV-positive Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2000-05; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
To determine the effectiveness of fixed dose(s) of NESP, administered once every other week, in the treatment of anemia in subjects with CRI | entire study - 24 weeks

SECONDARY OUTCOMES:
To assess the safety and tolerability of chronic NESP therapy | entire study - 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Suranyi MG, Lindberg JS, Navarro J, Elias C, Brenner RM, Walker R. Treatment of anemia with darbepoetin alfa administered de novo once every other week in chronic kidney disease. Am J Nephrol. 2003 Mar-Apr;23(2):106-11. doi: 10.1159/000068041. PMID 12481149
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_33_NESP_990151.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com